CLINICAL TRIAL: NCT00756678
Title: Efficacy and Acceptability of Two Lubricant Eye Drops
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MA-OPT-08-001
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-09

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Carboxymethylcellulose and Glycerin
  Interventions: Drug: Lubricant Eye Drops (Optive™)
- 2 (Active Comparator): Polyethylene glycol 400
  Interventions: Drug: Lubricating Eye Drops (blink® Tears)

INTERVENTIONS:
Drug: Lubricant Eye Drops (Optive™) — 1 drop in both eyes as needed for 7 days'
  Other Names: Optive™
  Arms: 1
Drug: Lubricating Eye Drops (blink® Tears) — 1 drop in both eyes as needed for 7 days
  Other Names: blink® Tears
  Arms: 2

SUMMARY:
Efficacy and acceptability of two new artificial tears following two weeks of treatment in patients with dry eye. Patients will be randomized to 1 of 2 treatments for 7 days then crossover to the alternate treatment for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* At least 18 years of age
* Current use of artificial tears

Exclusion Criteria:

* Any uncontrolled systemic disease
* Pregnancy or planning a pregnancy
* Contact lens wear

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Chevy Chase, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients
Period: Overall Study
Arm/Group | All Patients
Started | 51
Completed | 50
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 51
Age, Customized [Number; unit: participants]
  <=40 years | 22
  Between 40 and 65 years | 24
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Frequency of Eye Drop Use Over 1 Week
Description: Mean frequency of eye drop use per day per patient during the cross-over period over 1 week. Eye drop use was captured on a daily tear diary that the patients completed. The greater the frequency of use, the more eye drops were required to manage the patient's dry eye symptoms.
Time Frame: 1 week
Population: Intent to Treat; defined as all randomized (started study) patients. Of the 51 patients that were randomized, data for 50 patients were evaluated for this outcome measure
Measure: Mean (Standard Deviation); unit: Use per day
Groups:
- Lubricant Eye Drops (Optive™): Lubricant Eye Drops (Optive™)
- Lubricant Eye Drops (Blink® Tears): Lubricant Eye Drops(blink® Tears)
Arm/Group | Lubricant Eye Drops (Optive™) | Lubricant Eye Drops (Blink® Tears)
Number analyzed (Participants) | 50 | 50
Use per day | 1.76 (0.89921) | 1.66 (0.94459)

2. Secondary Outcome: Change From Baseline in Dry Eye Disease Comfort Assessment Score on Day 16
Description: Mean change from baseline in Dry Eye Disease Comfort Assessment Score at Day 16. The Dry Eye Disease Comfort Assessment consists of one question asking the patient to rate their current overall discomfort from their dry eye symptoms on a scale of 0 to 10 (0 equals No Discomfort; 10 equals Intolerable). The greater the negative number change from baseline, the greater the improvement in comfort.
Time Frame: Baseline, Day 16
Population: Intent to Treat; defined as all randomized (started study) patients. Of the 51 randomized patients, data from 49 patients were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lubricant Eye Drops (Optive™) | Lubricant Eye Drops (Blink® Tears)
Number analyzed (Participants) | 49 | 49
Scores on a scale
  Baseline | 4.65 (1.843) | 4.62 (1.839)
  Day 16 | -1.41 (2.010) | -1.47 (1.905)

3. Secondary Outcome: Percentage of Positive Patient Responses to Subject Acceptability Questionnaire on Day 16
Description: Percentage of patients who responded "Strongly Agree" and "Agree" to Subject Acceptability Questionnaire Question 1: Overall Liked. The Subject Acceptability Questionnaire consists of 11 multiple choice questions assessing how the patients feel about the eye drops received. The 5 possible responses to the questionnaire are "Strongly Agree", "Agree", "Neither Agree or Disagree", "Disagree" and "Strongly Disagree".
Time Frame: Day 16
Population: Intent to treat; defined as all randomized (started study)patients. Of the 51 randomized patients, data for 50 patients were evaluated for this outcome measure
Measure: Number; unit: Percentage of Patients
Arm/Group | Lubricant Eye Drops (Optive™) | Lubricant Eye Drops (Blink® Tears)
Number analyzed (Participants) | 50 | 50
Percentage of Patients | 86 | 78

4. Secondary Outcome: Number of Patients With Positive Responses to Subject Preference Questionnaire on Day 16
Description: Number of patients who marked that either Week 1 study product was more soothing or Week 2 study product was more soothing to the Overall Comfort Preference Questionnaire on Day 16 of the cross-over period. The Subject Preference Questionnaire consists of 4 questions related to comfort, soothing, blurring and purchase preference comparing treatments received during Week 1 versus Week 2.
Time Frame: Day 16
Population: Intent to Treat; defined as all randomized (started study) patients.
Measure: Number; unit: Number of patients
Arm/Group | Lubricant Eye Drops (Optive™) | Lubricant Eye Drops (Blink® Tears)
Number analyzed (Participants) | 51 | 51
Number of patients | 16 | 22

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.